CLINICAL TRIAL: NCT02898649
Title: Safety and Efficacy of Irreversible Electroporation for Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0150
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IRE (Experimental): The intervention group
  Interventions: Device: Irreversible electroporation

INTERVENTIONS:
Device: Irreversible electroporation — IRE is operated to tumor under laparotomy or CT-guided percutaneous approach. Unipolar (19G) or bipolar (16G) electrode probe is inserted to around tumor. After insertion of probe, short duration (70-90㎲) of electric current (25~45A) is generated by IRE device (NanoKnife IRE device, AngioDynamics, Queens bury, New York). It is possible to obtain a three-dimensional ablation zone using multiple electrode. IRE can cause apoptosis of tumor cells, without adjacent tissue damage.

SUMMARY:
Pancreatic cancer is 5th leading cause of cancer-related death in Korea. It has a dismal prognosis with very low 5-year survival rate, about 5%. Only 10% of pancreatic cancer patients is diagnosed in operable status. So, most of patients could not be treated with curative resection.

Locally advanced pancreatic cancer (LAPC) is defined by defined as surgically unresectable due to vascular encasement (e.g. celiac trunk or superior mesenteric artery) by tumor, but have no evidence of distant metastases. In LAPC patients, systemic chemotherapy with/without radiotherapy was used as a standard therapy, but therapeutic response was very poor. Only less than 30% of patients showed treatment response, and median survival of LAPC patient was only 9 months. Thus, more effective treatment modality is needed for LAPC patients.

Irreversible electroporation (IRE) is a soft tissue ablation technique using ultra short but strong electrical fields to create permanent and hence lethal nanopores in the cell membrane, to disrupt the cellular homeostasis. IRE does not cause thermally induced necrosis and has tissue selectivity, so adjacent tissue or vascular structures can be preserved.

Several clinical trials using IRE were performed to liver, kidney or lung cancer patients. We will operate IRE procedure to LAPC patients who were previously received standard therapy but showed no response, using NanoKnife IRE device. We will investigate treatment response and safety of IRE.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed pancreatic cancer patients
* Locally advanced pancreatic cancer patients. Vascular encasement by tumor was noted in radiological evaluation (CT, MRI or PET-CT)
* Older than 19 years old and younger than 70 years old
* Previously treated with systemic chemotherapy or chemoradiotherapy due to locally advanced pancreatic cancer.

Exclusion Criteria:

* Patients with life-threatening systemic disease.
* Metastatic or borderline-resectable pancreatic cancer patients
* Patients with seizure history
* Patients with arrythmia or heart failure
* Recent history of myocardial infarction (within 1 year)
* Patients who have implantable electronic devices. (e.g. pacemaker, defibrillator)
* Patients who have metal devices (e.g. metal stent) around tumor.
* Coagulopathy patients.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | from 1 month to 3 month
  Overall survival is calculated from the date of informed consent acquisition until the date of death.
Safety (frequency of procedure-related complication and death) | from 1 month to 3 month
  Safety is evaluated by the frequency of procedure-related complication and death.

SECONDARY OUTCOMES:
Time to progression | within 1 year
Tumor control | within 1 year
Pain control | within 1 year
Change in CA 19-9 | within 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university of medical center, Seoul, South Korea